CLINICAL TRIAL: NCT00488748
Title: Magnetic Seizure Therapy (MST) for the Treatment of Severe Mood Disorder
Brief Title: Magnetic Seizure Therapy (MST) for Severe Mood Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sarah Lisanby (Other)
Collaborators: Duke University (Other); University of Texas Southwestern Medical Center (Other); Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Sarah Lisanby, Professor and Chair, Department of Psychiatry and Behavioral Sciences, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00026868; Stanley Grant #05T656
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Depression
Keywords: MST; Magnetic Seizure Therapy; ECT; Electroconvulsive Therapy; Depression; Magnetic
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MST (Experimental): Magnetic Seizure Therapy (MST)
  Interventions: Device: Magstim Theta
- ECT (Active Comparator): Electroconvulsive Therapy (ECT)
  Interventions: Device: Thymatron

INTERVENTIONS:
Device: Thymatron — Right unilateral placement, 6x seizure threshold, 3 times per week until clinically appropriate to stop (approximately 2-6 weeks)
  Other Names: Thymatron, Electroconvulsive Therapy (ECT)
  Arms: ECT
Device: Magstim Theta — 100% power, vertex placement, 3 times per week, until clinically appropriate to stop (approximately 2-6 weeks)
  Other Names: Magstim Theta, Magnetic Seizure Therapy (MST)
  Arms: MST

SUMMARY:
This study will compare the clinical efficacy and side effects of Magnetic Seizure Therapy (MST) and Electroconvulsive Therapy (ECT) in patients currently experiencing a major depressive episode in the context of either unipolar or bipolar depression. The investigators will conduct a number of clinical and neuropsychological tests to assess clinical and cognitive response to treatment. The investigators hypothesize that:

1. MST and ECT will have similar antidepressant efficacy.
2. MST will have less post-treatment amnesia than ECT as reflected in primary measures of anterograde and retrograde amnesia following the acute treatment phase.
3. At follow up, MST will show a lesser degree of persisting deficit in measures of retrograde amnesia than ECT.

DETAILED DESCRIPTION:
The purpose of this study is to compare the clinical efficacy and side effects of Magnetic Seizure Therapy (MST) and Electroconvulsive Therapy (ECT) in patients currently experiencing a major depressive episode in the context of either unipolar or bipolar depression. ECT is known to be highly effective in treating depression, but it can have some adverse cognitive side effects. MST is a new form of convulsive therapy that is being developed as a means of improving the side effect profile of ECT so that more patients may benefit without suffering significant detrimental effects on cognition.

Both ECT and MST cause a seizure, but they do so in different ways. In ECT, an electrical stimulator is used to pass an electrical current between two electrodes placed on the person's head, which causes some electricity to go through the brain and cause a seizure. In MST, a magnetic stimulator is used to pass a magnetic field to the brain, which then creates a small electrical field in the brain that causes a seizure.

In addition to the treatment sessions, this study will involve a number of assessments at different timepoints that are used to evaluate the person's antidepressant response and the physical and cognitive side effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Clinical diagnosis of major depressive episode, in the context of unipolar or bipolar disorder
* Use of effective method of birth control for women of child-bearing capacity
* Willing and capable to provide informed consent
* Convulsive therapy clinically indicated
* Hamilton Rating Scale for Depression (HRSD24) ≥ 20

Exclusion Criteria:

* Current unstable or serious medical condition, or any comorbid medical condition that substantially increases the risks of ECT (such as acute myocardial infarction, space occupying brain lesion or other cause of increased intracranial pressure, unstable aneurysm or vascular malformation, poorly controlled diabetes mellitus, carcinoma, renal failure, hepatic failure)
* Pregnancy
* History of neurological disorder, epilepsy, stroke, brain surgery, metal in the head, history of known structural brain lesion
* Presence of devices that may be affected by MST (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Breast-feeding
* History of head trauma with loss of consciousness for greater than 5 minutes
* History of schizophrenia, schizoaffective disorder, or rapid cycling bipolar disorder
* Vagus nerve stimulator implanted
* History of substance abuse or dependence in past 3 months
* Failure to respond to an adequate course of ECT in the current depressive episode
* History of ECT in the past 6 months and/or failure to respond to an adequate trial of ECT lifetime
* Presence of intracardiac lines

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Clinical improvement (Hamilton Rating Scale for Depression) | After each treatment and at follow-ups up to 6 months after the treatment course

SECONDARY OUTCOMES:
Clinical improvement (Inventory of Depressive Symptomatology - Clinician-Rated) | Before and after treatment course, and at follow-ups up to 6 months after the treatment course

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H. Lisanby, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Lisanby SH, Luber B, Schlaepfer TE, Sackeim HA. Safety and feasibility of magnetic seizure therapy (MST) in major depression: randomized within-subject comparison with electroconvulsive therapy. Neuropsychopharmacology. 2003 Oct;28(10):1852-65. doi: 10.1038/sj.npp.1300229. PMID 12865903
- [Background] Kosel M, Frick C, Lisanby SH, Fisch HU, Schlaepfer TE. Magnetic seizure therapy improves mood in refractory major depression. Neuropsychopharmacology. 2003 Nov;28(11):2045-8. doi: 10.1038/sj.npp.1300293. PMID 12942146
- [Derived] Deng ZD, Luber B, McClintock SM, Weiner RD, Husain MM, Lisanby SH. Clinical Outcomes of Magnetic Seizure Therapy vs Electroconvulsive Therapy for Major Depressive Episode: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Mar 1;81(3):240-249. doi: 10.1001/jamapsychiatry.2023.4599. PMID 38055283
- [Derived] Jiang J, Zhang C, Li C, Chen Z, Cao X, Wang H, Li W, Wang J. Magnetic seizure therapy for treatment-resistant depression. Cochrane Database Syst Rev. 2021 Jun 16;6(6):CD013528. doi: 10.1002/14651858.CD013528.pub2. PMID 34131914
- See also: National Institute of Mental Health - Depression — http://www.nimh.nih.gov/publicat/depression.cfm
- See also: Summary of MST study on Duke Health website — http://www.dukehealth.org/clinicaltrials/magnetic-seizure-therapy-mst-for-the-treatment-of-severe-mood-disorder